CLINICAL TRIAL: NCT07022457
Title: UK ENcorafenib and BInimetinib Real-world Study in Melanoma (UK-EnBiRiM): A Prospective Observational Real-world App-based Study to Explore HRQoL Outcomes, of Adults With Metastatic Cutaneous BRAF V600 Mutation-positive Melanoma, Initiated on Combination Encorafenib and Binimetinib Therapy in the UK
Brief Title: UK ENcorafenib and BInimetinib Real-world Study in Melanoma
Acronym: UK-EnBiRiM
Status: Recruiting | Type: Observational
Sponsor: Pierre Fabre Ltd (Industry)
Collaborators: Vitaccess Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 5126-10-2024
Record Dates: First submitted 2025-05-16; First posted 2025-06-15 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Melanoma, BRAF V600 Mutation Positive
Keywords: Melanoma; BRAF V600; HRQoL; PROs; Encorafenib; Binimetinib; Real-World; prospective
MeSH Terms: conditions — Melanoma | interventions — encorafenib; binimetinib

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- UK-EnBiRiM study participants: Adult patients diagnosed with metastatic cutaneous BRAF V600 mutation-positive melanoma and assigned to receive encorafenib plus binimetinib as second-line treatment for metastatic melanoma, as per current Summary of Product Characteristics.
  Interventions: Biological: Encorafenib + Binimetinib

INTERVENTIONS:
Biological: Encorafenib + Binimetinib — Participants will have received a clinical decision to begin encorafenib plus binimetinib treatment as a second-line treatment for metastatic melanoma, in accordance with current Summary of Product Characteristics

SUMMARY:
This is a prospective longitudinal multi-centre observational study conducted in the United Kingdom, in patients with metastatic cutaneous BRAF V600 mutation-positive melanoma assigned to receive encorafenib and binimetinib. The aim of this study is to learn about how encorafenib and binimetinib perform, patients' experiences of using them, and how they might affect patient's quality of life, in the real world, when these treatments are prescribed by doctors instead of in a clinical trial. Participants will complete electronic data entry via questionnaires over a 24-month period. Site research teams will also complete electronic data entry using participants' medical records over a 24-month period.

DETAILED DESCRIPTION:
This longitudinal study will collect real-world clinical outcomes and patient-reported outcomes (PRO) data for patients receiving encorafenib plus binimetinib. The results from the study will be summarized descriptively to describe the impact of encorafenib plus binimetinib in the UK real-world setting.

The COLUMBUS trial has demonstrated the efficacy and safety profile of encorafenib plus binimetinib in patients with advanced melanoma with a BRAFV600 mutation; the 7-year analysis of this study is currently available. Real-world studies can reach broader patient populations than are typical of clinical trials, and also provide unique insights, such as real-life challenges faced by patients, the impact of a disease on productivity, and daily disease management. Given the importance of patient health-related quality of life (HRQoL) data in melanoma treatment and the potential value of real-world evidence (RWE), Pierre Fabre wishes to complement the clinical and HRQoL outcomes demonstrated for encorafenib plus binimetinib in the COLUMBUS trial with patient-reported outcomes (PROs) data from a real-world study.

The source population will be patients being treated for melanoma in National Health Service (NHS) England secondary care centers at the time of study enrolment. Approximately 8 study sites will be selected from the available secondary care centers, based on clinical experience with encorafenib plus binimetinib, research capacity, and willingness to take part.

Patients who are interested in participating in the study will be able to download the Vitaccess Real™ application either during their consultation at the site or at their own convenience. After completing the in-application informed consent process, they will be able to begin data entry via the application. Site research teams will complete an electronic case report form (eCRF) for each participant at baseline, using data from the participant's electronic medical record (EMR). For analysis purposes, data from the eCRF will be linked to the participant-reported data using the participant's assigned unique ID and PIN number.

ELIGIBILITY:
Inclusion criteria:

* Aged 18 years or older
* Willing and capable of providing written informed consent
* Access to a smartphone
* Diagnosis of metastatic cutaneous melanoma with presence of BRAF V600 mutation in tumour tissue prior to enrolment
* Clinical decision has been made to begin encorafenib plus binimetinib treatment in accordance with current Summary of Product Characteristics
* Encorafenib plus binimetinib to be prescribed as second-line treatment for BRAF V600-mutant metastatic melanoma

Exclusion criteria:

* Patients receiving systemic treatment for any tumours other than melanoma
* Patients participating in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with metastatic cutaneous BRAF V600 mutation-positive melanoma and assigned to receive encorafenib plus binimetinib as second-line treatment for metastatic melanoma, as per current Summary of Product Characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2028-01-13 (Estimated); Study Completion 2028-01-13 (Estimated)

PRIMARY OUTCOMES:
Describe the change from baseline over 24 months of FACT-Melanoma (FACT-M) scores of patients initiated on encorafenib plus binimetinib | Every eight weeks (±7 days) from baseline for first 6 months; every 3 months (±7 days) thereafter for the remaining 18 months (24 months total)
  FACT-M instrument data reported by patients via the Quality of Life - Melanoma in the UK (QOL-MUK) platform ("Impact of melanoma on well-being" survey). The FACT-M contains 24-items reported on a 5-point Likert-type scale ("Not at all", "A little bit", "Somewhat", "Quite a bit", and "very much"). The outcome measure contains the 3 QoL domains; 20 items relate to physical well-being, 3 to emotional well-being, and 1 to social well-being. The higher the score, the better the quality of life (QOL).

SECONDARY OUTCOMES:
Describe patient demographics | Once, at baseline
  Assessed using demographic data reported by participants via the QOL-MUK platform (including; month and year of birth, sex and ethnicity).
Describe patient baseline clinical characteristics | Once, at baseline
  Assessed using electronic medical record (EMR) data reported by healthcare professionals (HCPs) ("Disease history", "Statuses" and "Treatment history" surveys).
Describe median duration of treatment with encorafenib and binimetinib | Every three months (±7 days) for 24 months, starting three months from baseline
  Assessed using electronic medical record (EMR) data reported by healthcare professionals (HCPs) ("Treatment history" and "Treatment status" surveys).
Describe change from baseline over 24 months of EQ-5D-5L scores of patients receiving encorafenib plus binimetinib | Every eight weeks (±7 days) from baseline for first six months; every three months (±7 days) for the remaining 18 months (24 months total)
  EQ-5D-5L instrument data reported by patients via the QOL-MUK platform ("General health" survey). The instrument comprises two parts. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with 5 levels (1 - no problems, 2 - slight problems, 3 - moderate problems, 4 - severe problems, and 5 - extreme problems). The digits for 5 dimensions can be combined in a 5-digit number describing the health state of the person.
Describe changes in patient self-reported symptom severity over 24 months using the Patient Global Impression of Severity (PGI-S) | Every eight weeks (±7 days) from baseline for first six months; every three months (±7 days) for the remaining 18 months (24 months total)
  PGI-S instrument data will be reported by patients via the QOL-MUK platform ("Symptom severity" survey). This is a generic instrument used to assess self-perceived severity of a specific condition, with the following response options: None, Mild, Moderate, Severe, Very Severe.
Describe the median time from baseline to definitive 10% deterioration of the FACT-M scores of patients receiving encorafenib plus binimetinib using Kaplan-Meier analysis | Every eight weeks (±7 days) from baseline for first six months; every three months (±7 days) for the remaining 18 months (24 months total)
  FACT-M instrument data reported by patients via the QOL-MUK platform ("Impact of melanoma on well-being" survey). A 10% deterioration is defined as a deterioration of at least 10% in total FACT-M score. The total FACT-M score ranges from 0 to 172. The higher the FACT-M score, the better the QOL.
Describe the median time from baseline to definitive 10% deterioration of the EQ-5D-5L scores of patients receiving encorafenib plus binimetinib using Kaplan-Meier analysis | Every eight weeks (±7 days) from baseline for first six months; every three months (±7 days) for the remaining 18 months (24 months total)
  EQ-5D-5L instrument data will be reported by patients via the QOL-MUK platform ("General health" survey). A 10% deterioration is defined as a deterioration of at least 10% in the utility index score for EQ-5D-5L. EQ-5D-5L utility index scores range from 0 to 1; higher index scores indicate a higher health utility.
Describe reasons why encorafenib plus binimetinib treatment may be discontinued | Every three months (±7 days) for 24 months, starting three months from baseline
  Assessed using electronic medical record (EMR) data reported by healthcare professionals (HCPs) ("Treatment status" survey).
Describe real-world progression-free survival (PFS) and overall survival (OS) of patients receiving encorafenib plus binimetinib using Kaplan-Meier analysis | Every three months (±7 days) for 24 months, starting three months from baseline
  Assessed using electronic medical record (EMR) data reported by healthcare professionals (HCPs) ("Clinical outcomes" survey).
Describe the presence of melanoma brain metastases (MBM) at the beginning of study and the development and/or progression of MBM in patients receiving encorafenib plus binimetinib | Every three months (±7 days) for 24 months, starting three months from baseline
  Assessed using electronic medical record (EMR) data reported by healthcare professionals (HCPs) ("Clinical outcomes" survey), specifically whether melanoma has metastasized to brain since previous assessment; if new MBM, date of metastasis; if existing MBM, whether intracranial progression; if yes, date of intracranial progression.
Describe adverse events (AEs) experienced by patients receiving encorafenib plus binimetinib | Within 24 hours of becoming aware of AEs
  This will be assessed via the contents of Pierre Fabre solicited AE collection form, including type of AE and grade/severity.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Furness, MBBS, MRCP, PhD, Principal Investigator — Royal Marsden NHS Foundation Trust; Tarandeep Singh Matharu, MPharm, PgCert, Study Director — Pierre Fabre Limited
Locations (7):
- United Kingdom (7):
  - Southend University Hospital, Westcliff-on-Sea, Essex
  - Queen Elizabeth Hospital, Birmingham
  - Addenbrookes Hospital, Cambridge
  - University Hospital Coventry and Warwickshire, Coventry
  - Royal Marsden Hospital, London
  - Royal Preston Hospital, Preston
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No